CLINICAL TRIAL: NCT02756585
Title: Computed Tomography Perfusion in Patients With Severe Head Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP TBI
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2016-04

CONDITIONS: Brain Injuries
Keywords: computed tomography; perfusion imaging; brain death; traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Brain Death; Brain Injuries, Traumatic | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ct perfusion (Other): All participants will undergo the imaging protocol with CTP of head at the time of initial diagnostic imaging upon hospital arrival.
  Interventions: Radiation: ct perfusion

INTERVENTIONS:
Radiation: ct perfusion — computed tomography perfusion of the head

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of post-injury hospitalization, disability, and death worldwide. In Nova Scotia, approximately 50% of major trauma reported is head trauma. TBI is predicted to be the most common and expensive neurological condition in Canada through the year 2031.

Families and medical teams must often decide on the appropriate level of care for patients with severe TBI and frequently need to consider withdrawal of life support measures. These decisions have implications for patients with severe TBI, costs to the health care system, and rates of organ donation.

A reliable method for neurological evaluation at the time of the patient's arrival to the hospital is important, because it is possible that many patients with severe TBI already have permanent brain damage. Assessing this brain damage with clinical tests is difficult because of the nature of patients' injuries and the sedative medication they receive at the time of their hospital admission. Current standard imaging technique for these patients is severely limited in the assessment of the extent and severity of the brain damage.

Advanced diagnostic imaging, called Computed Tomography Perfusion (CTP), can help detect permanent brain damage. However, CTP of the head is not currently done for patients with severe TBI when they arrive at the hospital. The investigators want to test whether CTP of the head can detect permanent brain damage among patients with severe TBI.

DETAILED DESCRIPTION:
To demonstrate that CTP is useful for assessing patients with severe TBI, the investigators will conduct a large study at multiple hospitals across Canada. Before conducting the large study, the investigators need to make sure that it is feasible to add CTP of the head to the routine imaging that patients with severe TBI undergo at the time of their arrival at the hospital. The current study is a pilot study to test the feasibility of adding CTP imaging of the head to the routine imaging protocol for patients with severe TBI at the time of their hospital admission. The proposed feasibility study will help determine how many participants the investigators need for the larger study to attain a significant result and whether the investigators need to modify the investigators study methods.

Participants will undergo the imaging protocol with CTP of head at the time of initial diagnostic imaging upon hospital arrival. Non-contrast CT (NCCT) of the head will be performed as part of current imaging protocol for severe TBI patients. At the time of the NCCT, participants will undergo whole-brain CTP protocol, ensuring coverage of the entire brainstem. A total of 40 mL of nonionic iodinated contrast media will be injected. Images will be acquired according to the investigators previously published imaging protocol. Cerebral blood flow (CBF) and cerebral blood volume (CBV) images from the CTP will be qualitatively assessed for the presence or absence of a matched decrease of CBF and CBV in the brainstem. CTP will be assessed independently by two radiologists blinded from each other. If disagreements arise, they will be resolved by discussion.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* severe head injury with Glasgow Coma Scale score ≤ 8 after initial resuscitation
* on mechanical respiratory support at the time of imaging

Exclusion Criteria:

* known to be pregnant
* any known contraindication to CT contrast agent, such as an allergy or anaphylactic reaction
* known end-stage renal disease (on chronic dialysis or to be expected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
death | until hospital discharge, up to 1 year
  the death of the participant due to any cause at discharge

SECONDARY OUTCOMES:
recruitment rate | through study completion, up to 2 years
  Number of potential participants approached who agreed to participate

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II Health Sciences Centre-Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shankar JJ, Vandorpe R. CT perfusion for confirmation of brain death. AJNR Am J Neuroradiol. 2013 Jun-Jul;34(6):1175-9. doi: 10.3174/ajnr.A3376. Epub 2012 Dec 28. PMID 23275594